CLINICAL TRIAL: NCT06762301
Title: The Effect of Sexual Education-Counseling According to PLISSIT Model of Couples' Sexual Functions During Pregnancy and Postpartum
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Özlem BAKAN DEMİREL, Phd candidate, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARMARAU-SBE-OBD-01
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy; Postpartum Period; Sexual Dysfunction; PLISSIT Model; Sexual Counselling
Keywords: pregnancy; postpartum period; sexual dysfunction; PLISSIT model; sexual counselling
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participant Group (Experimental): After the initial evaluation, pregnant women who will be included in the study group will be given an appointment for 1 week later, they will be asked to come with their partners and couples will be given sexual education and counseling in line with the PLISSIT model.
  After the initial evaluation, couples will be interviewed in the 1st, 2nd and 3rd trimesters, their sexuality since the previous evaluation according to the PLISSIT model, their problems, if any, will be discussed and short counseling will be given if necessary.
  In the first 4 weeks after delivery, couples in the study group will receive sexual education and counseling for the postpartum period in line with the PLISSIT model.
  They will be interviewed at the 3rd and 6th month after delivery and their postpartum sexuality and problems, if any, will be discussed and the sexual functions of the couples for the last 4 weeks will be evaluated.
  Interventions: Behavioral: sexual education and counseling
- Control Group (Other): Routine clinical care
  Interventions: Other: Routine clinical care

INTERVENTIONS:
Behavioral: sexual education and counseling — After the initial evaluation, pregnant women who will be included in the study group will be given an appointment for 1 week later, they will be asked to come with their partners and couples will be given sexual education and counseling in line with the PLISSIT model. After the initial evaluation, couples will be interviewed in the 1st, 2nd and 3rd trimesters, their sexuality since the previous evaluation according to the PLISSIT model, their problems, if any, will be discussed and short counseling will be given if necessary. In the first 4 weeks after delivery, couples in the study group will receive sexual education and counseling for the postpartum period in line with the PLISSIT model. They will be interviewed at the 3rd and 6th month after delivery and their postpartum sexuality and problems, if any, will be discussed and the sexual functions of the couples for the last 4 weeks will be evaluated.
  Arms: Participant Group
Other: Routine clinical care — Control Group
  Arms: Control Group

SUMMARY:
Sexuality is a natural part of human life at every stage of life. It is a multidimensional phenomenon influenced by biological, psychological, social, interpersonal and cultural factors. Pregnancy is an extremely important process that occurs as a result of a sexual relationship and affects the lives of the woman and the couple.

Many studies in the literature clearly show that sexual life is affected during pregnancy and postpartum period. In this context, it is stated that sexual health assessment, sexual education and counseling in pregnant/couples can be addressed in the early stages of pregnancy to reduce the anxiety of couples and the likelihood of sexual problems. It is important to evaluate sexual health during pregnancy and postpartum and to provide counseling and support in line with the results. In order to evaluate pregnancy and postpartum processes appropriately, the sexual history of women/couples should be defined. Therefore, it is important to learn the pre-pregnancy history of women/couples regarding their sexual activities and current sexual functions, to determine whether they experience sexual dysfunction during pregnancy or postpartum, and to examine its role in pregnancy and postpartum period, if any.

DETAILED DESCRIPTION:
Many studies in the literature clearly show that sexual life is affected during pregnancy and postpartum period. In this context, it is stated that sexual health assessment, sexual education and counseling in pregnant/couples can be addressed in the early stages of pregnancy to reduce the anxiety of couples and the likelihood of sexual problems. It is important to evaluate sexual health during pregnancy and postpartum and to provide counseling and support in line with the results. In order to evaluate pregnancy and postpartum processes appropriately, the sexual history of women/couples should be defined. Therefore, it is important to learn the pre-pregnancy history of women/couples regarding their sexual activities and current sexual functions, to determine whether they experience sexual dysfunction during pregnancy or postpartum, and to examine its role in pregnancy and postpartum period, if any.In this context, talking to couples about their sexuality and providing sexual health counseling appropriate to their needs provides an opportunity to develop safe sexual health behaviors. In this process, the aim of nurses is to strengthen the sexual health of couples, encourage them to express their sexual problems, determine the causes and characteristics of sexual problems, and make interventions for the problems identified. The nurse can plan and carry out preventive interventions for the sexual health of couples, improve the ability to express sexual life, counsel and refer for early diagnosis and treatment of existing problems. It is recommended to use a model that will be useful in the training and counseling services provided by nurses and it is stated that it will increase the effectiveness of the service provided.It is emphasized that the PLISSIT model is a useful tool for nurses on sexuality and sexual health. The PLISSIT model supports the counseling role by assessing the individual in collaboration, understanding and respecting their decisions. By using the first three phases of this model, which can be applied at any time and in different situations, 80-90% of sexual problems can be solved on average. Recent studies in the literature with this model show that the training and counseling provided according to the models have positive effects on sexual problems.

In the studies conducted, it was observed that sexual education and counseling processes did not include pregnant women and their partners, and there were no studies evaluating the long-term effects on the sexual lives of couples. In this study, it was aimed to determine the effect of sexual education-counseling given to couples with sexual dysfunction in the preconceptional period in accordance with the PLISSIT model on their sexual functions during pregnancy and postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* For a pregnant woman;
* A woman who had just received the result of a pregnancy test and was referred to the family health center due to a positive pregnancy,
* Who wants the pregnancy to continue,
* In the first 6-8 gh. of gestation,
* FSFI cut-off value for pre/conceptional period with a total score ≤26.55,
* The one with a single, healthy fetus,
* Has a sexual partner and has an active sexual life,
* For the pregnant woman and her partner/partner;
* Educated enough to understand what they read and answer questions,
* Do not have chronic diseases that may affect sexual health (cancer, diabetes, hypertension, hypercholesterolemia, heart disease, atherosclerosis, chronic pulmonary and hepatic diseases, chronic renal failure, mental disorder, etc.) or continuous drug use (antihypertensive, diuretic, lipid-lowering agent, H2 receptor antagonist, antihistamine, anticholinergic, chemotherapeutic agent, anticonvulsant, antidepressant, antipsychotic, narcotic, sedative, etc.) and
* Pregnant women and their spouses who volunteered to participate in the study

Exclusion Criteria:

* Not planning to continue the pregnancy / planning to terminate the pregnancy,

  * Who has completed the first trimester of pregnancy,
  * FSFI cut-off value for pre/conceptional period with a total score >26.55
  * No active sex life,
  * With language problems,
  * Not educated enough to understand what they read and answer questions,
  * Chronic illness or medication that may affect sexuality,
  * Those who did not want to participate in the study and
  * Pregnant women and their partners who wanted to leave the study voluntarily at any stage of the study / who felt uncomfortable with the questions asked during the study, or who discontinued the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) | 15 Months
  According to the Female Sexual Function Index (FSFI) cut-off value to be applied to each sampled pregnant woman at the first encounter, pregnant women with a total score ≤26.55, that is, pregnant women with sexual dysfunction, will be identified.
The International Erectile Function Evaluation Form (IIEF) | 15 Months
  The International Erectile Function Evaluation Form (IIEF) is evaluated in 5 categories in terms of erectile function. These are; severe erectile dysfunction (ED) score (6-10), moderate ED score (11-16), moderate-mild ED score (17-21), mild ED score (22-25), no ED (26-30) (Cappelleri et al., 1999). The scores that can be obtained as a result of IIEF evaluation are between 5-75. Cut-off value is not specified.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No